CLINICAL TRIAL: NCT05360355
Title: Flap Fenestration and Facial Organ Fabrication Guided By Intraoperative Indocyanine Green Angiography in Total Facial Restoration
Brief Title: Flap Fenestration and Facial Organ Fabrication Guided by ICGA
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Tao Zan, MD, Ph.D, Clinical professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: ICGA Guided Flap Fenestration
Record Dates: First submitted 2022-04-19; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Surgery
Keywords: Total facial restoration, Indocyanine green angiography, Flap fenestration, Facial organ fabrication, Flap surgery, Case series

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- patients undergone total face reconstruction and intraoperative indocyanine green angiography: This clinical study enrolled 10 patients treated with total face reconstruction and intraoperative indocyanine green angiography from Jun 2018 to Jun 2021.
  Interventions: Procedure: total face reconstruction surgery and intraoperative indocyanine green angiography

INTERVENTIONS:
Procedure: total face reconstruction surgery and intraoperative indocyanine green angiography — Patients with total facial scarring following burn injury were treated with monoblock pre-expanded prefabricated flaps for total face restoration. The opening of nostrils, oral and palpebral orifices, together with organ fabrication, were conducted under the guidance of intraoperative ICGA for hemodynamic evaluation.

SUMMARY:
In this retrospective study, patients with severe head and neck deformity were treated with monoblock pre-expanded prefabricated flaps for total face restoration. The opening of nostrils, oral and palpebral orifices, together with organ fabrication, were conducted under the guidance of intraoperative ICGA for hemodynamic evaluation. The hemodynamic analysis of flap perfusion before and after fenestration. Postoperative follow-up including vascular crisis, infection, flap necrosis and patients' aesthetic and functional recovery.

DETAILED DESCRIPTION:
The study included patients with severe head and neck deformity treated by our reconstructive team from Jun 2018 to Jun 2021, with monoblock pre-expanded flaps from the anterior chest, abdomen or back. For flap harvested from the chest, flap prefabrication was conducted in the first stage. In brief, the full length of the descending branch of the lateral circumflex femoral artery, vein and surrounding fascia were harvested and transferred as a free vascular carrier to the subcutaneous space on the anterior thoracic region. The pedicle vessels were anastomosed to the superior thyroid or facial vessels. A rectangular tissue expander was placed underneath the vascular carrier for expansion. In the second stage, the prefabricated flap was transferred to the pedicle vessel to replace the facial defects. Notably, dominant perforators were detected preoperatively and preserved during flap harvest for potential vascular anastomosis. For flaps from the abdomen and back, flaps were harvested as multi-pedicle free flaps. Exclusion criteria included severe liver, kidney or lung insufficiency, and allergy to iodine products.

Upon flap transfer to the face, a 2 mL bolus of ICG (2.5mg/mL) was administrated intravenously and the fluorescence signals were detected by a SPY imaging system (Novadaq Technologies, Inc., Canada). The course of each nourishing vessels and their respective perfusion territory were assessed. During flap fenestration, the opening of oral orifice was given the highest priority, followed by nostrils and palpebral orifices. If the region intended for flap fenestration was well perfused and did not contain major communicating branches or the penetration point of perforators, orifices would be opened directly. In the event of insufficient blood supply, additional vascular anastomosis would be considered for perfusion augmentation, and ICGA would be reconducted for evaluation.

The hemodynamic analysis of flaps was performed before and after fenestration using the incorporated SPY-Q software. The patients' aesthetic and functional recovery were evaluated, as well as postoperative complications including vascular crisis, infection, and flap necrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative facial soft tissue deformities/defects of type III and IV
2. Patients treated with monoblock pre-expanded prefabricated flaps for total face restoration.
3. Agreed and able to cooperate with the follow-ups, with signed informed consent form or audio recorded informed consent.

Exclusion Criteria:

1. Patients with severe liver, kidney or lung insufficiency, and allergy to iodine products
2. Patients with mental illness, reduced cognitive capacity, unable to consent and unable to cooperate.
3. Minor patients without legal guardian.
4. Not willing to participate; informed consent form not signed.

Ages: 4 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: This clinical study will include patients treated with total face restoration surgeries and intraoperative indocyanine green angiography from Jun 2018 to Jun 2021. It is estimated that about 10 patients will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The arterial infusion rate of flap before flap fenestration | 10 minutes
  The flap perfusion before flap fenestration was recorded by indocyanine green angiography (SPY imaging system, Novadaq Technologies Inc, Canada). The arterial infusion rate of flap perfusion before flap fenestration was calculated using the incorporated SPY-Q software.
The arterial infusion rate of flap after flap fenestration | 10 minutes
  The flap perfusion after flap fenestration was recorded by indocyanine green angiography (SPY imaging system, Novadaq Technologies Inc, Canada). The arterial infusion rate of flap perfusion after flap fenestration was calculated using the incorporated SPY-Q software.

SECONDARY OUTCOMES:
The occurrence rate of flap necrosis | 2 weeks post-operation
  The occurrence rate of flap necrosis was calculated at 2 weeks postoperatively. Flap necrosis was determined by three surgeons postoperatively. Necrosis includes epidermolysis, partial/superficial necrosis, and full-thickness necrosis. Partial/superficial necrosis is defined as loss of epidermis and partial loss of dermis with no subcutaneous tissue exposure/no requirement for debridement. Full-thickness necrosis is defined as loss of both epidermis and dermis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data are only available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Huang X, Li H, Gu S, Gao Y, Khoong Y, Liu Y, Luo S, Gu B, Li Q, Zan T. Intraoperative Indocyanine Green Angiography Facilitates Flap Fenestration and Facial Organ Fabrication in Total Facial Restoration. Plast Reconstr Surg. 2024 Jun 1;153(6):1416-1424. doi: 10.1097/PRS.0000000000010891. Epub 2023 Jun 28. PMID 37382913